CLINICAL TRIAL: NCT03365648
Title: A Randomized, Double-blinded, Parallel-group, Placebo-controlled Clinical Study of the Efficacy and Safety of an Oral Nutraceutical (Lertal®) as an add-on to Standard Therapy for Allergic Rhinoconjunctivitis in Pediatrics
Brief Title: Efficacy and Safety of Lertal® as an add-on to Standard Therapy for Allergic Rhinoconjunctivitis in Pediatrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NTC srl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LER 02-2017
Record Dates: First submitted 2017-11-22; First posted 2017-12-07 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Allergic Rhinoconjunctivitis
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: A randomized, double-blinded, parallel-group, placebo-controlled clinical study
Who Masked: Participant, Investigator
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lertal® + standard therapy (Experimental): Lertal® double-layer tablets (1 tab/day for 4 weeks) plus standard therapy (antihistamine)
  Interventions: Dietary Supplement: Lertal® + standard therapy
- Placebo + standard therapy (Placebo Comparator): Placebo tablets (1 tab/day for 4 weeks) plus standard therapy (antihistamine)
  Interventions: Other: Placebo + standard therapy

INTERVENTIONS:
Dietary Supplement: Lertal® + standard therapy — Lertal® is a novel food supplement. Each tablet contains the following active ingredients:
  * Quercetin 150 mg: a natural flavonoid that inhibits the release of histamine, leukotrienes, PGD2, IL (IL-6, IL-8, TNF-alpha).
  * Perilla frutescens 80 mg: A dry extract of the seeds containing rosmarinic acid, luteolin, apigenin and crysoeriol that inhibits the release of histamine and expression of interleukins (IL-6, TNF-alpha).
  * Vitamin D3 5 mcg (200 IU), which contributes to the normal function of the immune system.
  Standard therapy: antihistamine.
  Arms: Lertal® + standard therapy
Other: Placebo + standard therapy — Placebo tablet identical in appearance, size and taste to Lertal® tablets. Standard therapy: antihistamine.
  Standard therapy: antihistamine
  Arms: Placebo + standard therapy

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Lertal® as an add-on treatment for children affected by allergic rhinoconjunctivitis.

DETAILED DESCRIPTION:
Allergic rhinoconjunctivitis (AR) is a common chronic disorder in children, especially in developed countries. It is not characterized by nasal symptoms only (such as congestion and sneezing), but may also cause general complaints such as fatigue and cough. AR can also have detrimental effects on mood, sleep, social activities and scholastic performance.

Lertal® is a novel nutraceutical containing seed extracts from Perilla Frutescens, Quercetin extracted from Sophora japonica and Vitamin D3, all compounds that have demonstrated their ability to reduce allergy symptoms and the use of anti-allergy drugs in adults.

The aim of this randomized, double-blinded, parallel-group, placebo-controlled study is to evaluate the efficacy and safety of Lertal® as an add-on treatment for children affected by allergic rhinoconjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 to 12 years
* Male or female
* Diagnosis of allergic rhinoconjunctivitis
* Hypersensitivity to dust mites or pollen confirmed with skin-prick test (wheal and redness, ≥ 3 mm more extended than control) performed in the previous 12 months
* Total Symptoms Score (TSS) ≥ 15 and at least 1 for nasal congestion
* Written informed consent of patient and of parent or legal guardian

Exclusion Criteria:

* Uncontrolled asthma
* Secondary rhinitis to other causes
* Documented evidence of acute or chronic sinusitis
* Nasal polyps
* Chronic or intermittent use of inhaled, oral, intramuscular, intravenous or topical corticosteroids
* Use of leukotriene antagonists
* Continuous use of antihistamines
* Inadequate washout of drugs:

  * Systemic or intranasal corticosteroids: 1 month
  * Leukotriene antagonists: 1 month
  * Sodium cromoglycate: 2 weeks
  * Systemic or intranasal decongestants: 3 days
  * Cetirizine, fexofenadine, loratadine, desloratadine, hydroxyzine: 5-10 days
* Malformations of the nose, ear or throat
* Upper or lower respiratory tract infection in the last 2 weeks
* Participation in other clinical studies in the last month
* Documented hypersensitivity to the study product or its excipients
* Trip planned outside of the study area

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2018-07-04 (Actual); Study Completion 2018-11-13 (Actual)

PRIMARY OUTCOMES:
Total Symptom Score (TSS) scores | At Baseline and after Visit 4 (Week 4)
  Changes from baseline of Total Symptom Score (TSS) scores will be calculated after 4 weeks of treatment. The Total Symptoms score is a patient-reported evaluation of nine symptoms:
  * Nasal symptoms (Total Nasal Symptom Score): itching, sneezing, rhinorrhea, nasal congestion
  * Ocular symptoms (Total Ocular Symptom Score): itching, hyperemia of conjunctiva, tearing
  * Throat symptoms (Total Throat Symptom Score): itching, coughing
  With the help of their parents, patients will score symptoms on a 4-point scale: 0 = absent or irrelevant, 1 = mild, 2 = moderate, 3 = severe. Patients are asked to assign a score to the symptoms experienced in the last 12 hours and over the previous two weeks.
  The total symptom score is the sum of the scores of nasal symptoms, ocular symptoms and throat symptoms.
  The between-group analysis will be performed by means of a t-test for independent samples or analogous non-parametric test.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) score | At Baseline, after Visit 3 (Week 2) and after Visit 4 (Week 4)
  The patient will be asked to indicate overall system distress on a 100 mm Visual Analogue Scale (VAS) were 0 is equal to no discomfort and 100 the worst possible discomfort. Change from baseline of Visual Analogue Scale (VAS) score after 2 and 4 weeks of treatment. The between-group analysis will be performed using a t-test for independent samples or analogous nonparametric test.
Total Symptom Score (TSS) scores | At Baseline and after Visit 3 (Week 2)
  Change from baseline of Total Symptom Score (TSS) scores after 2 weeks of treatment. The Total Symptoms score is a patient-reported evaluation of nine symptoms:
  * Nasal symptoms (Total Nasal Symptom Score): itching, sneezing, rhinorrhea, nasal congestion
  * Ocular symptoms (Total Ocular Symptom Score): itching, hyperemia of conjunctiva, tearing
  * Throat symptoms (Total Throat Symptom Score): itching, coughing
  With the help of their parents, patients will score symptoms on a 4-point scale: 0 = absent or irrelevant, 1 = mild, 2 = moderate, 3 = severe. Patients are asked to assign a score to the symptoms experienced in the last 12 hours and over the previous two weeks.
  The total symptom score is the sum of the scores of nasal symptoms, ocular symptoms and throat symptoms.
  The between-group analysis will be performed by means of a t-test for independent samples or analogous non-parametric test.
Number of responders (30% reduction of TSS) | After Visit 3 (Week 2) and after Visit 4 (Week 4)
  Change from baseline of TSS score for each patient after 2 and 4 weeks of treatment will be classified as ≥ 30% and < 30%, thus defining responder and non-responder patients. Between-group differences will be tested by means of a Chi-square test with 2x2 contingency tables.
Time to maximum effect on Total Symptom Score (TSS) vs placebo | From baseline to Visit 6 (Week 16)
  Time to maximum effect on Total Symptom Score (TSS) vs placebo will be analysed by means of t-test for independent samples after logtransformation of the data or analogous non-parametric test. The Total Symptoms score is a patient-reported evaluation of nine symptoms:
  * Nasal symptoms (Total Nasal Symptom Score): itching, sneezing, rhinorrhea, nasal congestion
  * Ocular symptoms (Total Ocular Symptom Score): itching, hyperemia of conjunctiva, tearing
  * Throat symptoms (Total Throat Symptom Score): itching, coughing
  With the help of their parents, patients will score symptoms on a 4-point scale: 0 = absent or irrelevant, 1 = mild, 2 = moderate, 3 = severe. Patients are asked to assign a score to the symptoms experienced in the last 12 hours and over the previous two weeks.
  The total symptom score is the sum of the scores of nasal symptoms, ocular symptoms and throat symptoms.
Number of patients using rescue treatment | From baseline to Visit 6 (Week 16)
  Between-group differences in the number of patients using rescue treatment will be analyzed by means of a Chi-square test with 2x2 contingency tables.
Total Nasal Symptom Score (TNSS) | At Baseline, after Visit 3 (Week 2) and to Visit 4 (Week 4)
  The Total Nasal Symptom Score is a patient-reported evaluation of the following symptoms: itching, sneezing, rhinorrhea, nasal congestion. With the help of their parents, patients will score symptoms on a 4-point scale: 0 = absent or irrelevant, 1 = mild, 2 = moderate, 3 = severe. Patients are asked to assign a score to the symptoms experienced in the last 12 hours and over the previous two weeks.
  Changes from baseline in Total Nasal Symptom Score (TNSS) scores will be calculated after 2 and 4 weeks of treatment and between-group differences analyzed using a t-test for independent samples or analogous non-parametric test.
Total Ocular Symptom Score (TOSS) | At Baseline, after Visit 3 (Week 2) and to Visit 4 (Week 4)
  The Total Ocular Symptom Score is a patient-reported evaluation of the following symptoms: itching, hyperemia of conjunctiva, tearing. With the help of their parents, patients will score symptoms on a 4-point scale: 0 = absent or irrelevant, 1 = mild, 2 = moderate, 3 = severe. Patients are asked to assign a score to the symptoms experienced in the last 12 hours and over the previous two weeks.
  Changes from baseline in Total Ocular Symptom Score (TOSS) scores will be calculated after 2 and 4 weeks of treatment and between-group differences analyzed using a t-test for independent samples or analogous non-parametric test.
Total Throat Symptom Score (TTSS) | At Baseline, after Visit 3 (Week 2) and to Visit 4 (Week 4)
  The Total Throat Symptom Score is a patient-reported evaluation of the following symptoms: itching, coughing. With the help of their parents, patients will score symptoms on a 4-point scale: 0 = absent or irrelevant, 1 = mild, 2 = moderate, 3 = severe. Patients are asked to assign a score to the symptoms experienced in the last 12 hours and over the previous two weeks.
  Changes from baseline in Total Throat Symptom Score (TTSS) scores will be calculated after 2 and 4 weeks of treatment and between-group differences analyzed using a t-test for independent samples or analogous non-parametric test.
Number of patients symptom-free or with mild symptoms | From V3 (Week 2) to Visit 4 (Week 4)
  The number of patients with score for a single symptom ≤ 1 will be calculated and the between-group differences analyzed by means of a Chi-square test with 2xn contingency tables, where n represents the number of observations.
Number of exacerbations | From Visit 5 (Week 8) to Visit 6 (Week 16)
  Exacerbations are defined as the need of an antihistamine medication of any kind, at any dose and of any duration.
Intensity (mild, moderate, severe) of exacerbations | From Visit 5 (Week 8) to Visit 6 (Week 16)
  Exacerbations are defined as the need of an antihistamine medication of any kind, at any dose and of any duration.
Duration (number of days) of exacerbations | From Visit 5 (Week 8) to Visit 6 (Week 16)
  Exacerbations are defined as the need of an antihistamine medication of any kind, at any dose and of any duration.

OTHER OUTCOMES:
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) recorded throughout the study | From baseline to Visit 6 (Week 16)
  The incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) recorded throughout the study will be presented overall and by treatment group respectively.
Pediatric Rhinoconjunctivitis Quality of Life Questionnaire (PRQLQ) total score | At Baseline, at Visit 4 (Week 4) and at Visit 5 (Week 8) or Visit 6 (Week 16)
  The Pediatric Rhinoconjunctivitis Quality of Life Questionnaire consists of 23 questions in 5 domains (nasal symptoms, ocular symptoms, practical issues, limitation of activities, other symptoms), that are answered on a 7-point scale (0-6), where 0 represents the absence of problems and 6 the greatest symptom distress. Changes from baseline of the Pediatric Rhinoconjunctivitis Quality of Life Questionnaire total score will be calculated at Visit 4 (Week 4) and at Visit 5 (Week 8) or Visit 6 (Week16). An analysis of variance for repeated measures will be adopted, isolating the variability due to type of allergy, treatment group, time of observation and their interaction.

CONTACTS AND LOCATIONS:
Overall Officials: Gian Luigi Marseglia, Prof., Principal Investigator — Fondazione IRCCS Policlinico San Matteo di Pavia
Locations (17):
- Italy (17):
  - Fondazione IRCCS Policlinico San Matteo, Pavia, (PV)
  - Ospedale regionale San Salvatore - ASL 1 Avezzano Sulmona L'Aquila, L’Aquila, AQ
  - A.O.U. Consorziale "Policlinico Giovanni XXIII", Bari, BA
  - A.O.U. Consorziale "Policlinico-Giovanni XXIII", Bari, BA
  - A.O.U. Policlinico Vittorio Emanuele, Catania, CT
  - Istituto Giannina Gaslini, Genova, GE
  - P.O. San Giovanni di Dio - ASP di Crotone, Crotone, KR
  - A.O.U. Policlinico "G. Martino", Messina, ME
  - P.O. G. Salvini di Garbagnate Milanese - ASST Rhodense, Garbagnate Milanese, MI
  - Ospedale Civile di Legnano - ASST Ovest Milanese, Legnano, MI
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, MI
  - Ospedale San Carlo Borromeo - ASST Azienda Socio Sanitaria Territoriale Santi Paolo E Carlo, Milan, MI
  - Ospedale Città di Sesto San Giovanni - ASST Nord Milano, Sesto San Giovanni, MI
  - Ospedale di Polistena "Santa Maria degli Ungheresi" - ASP di Reggio Calabria, Polistena, RC
  - A.O.U. Policlinico Umberto I, Roma, RM
  - P.O. di Busto Arsizio - ASST Valle Olona, Busto Arsizio, VA
  - Az. Osp. Univ. dell'Università degli Studi della Campania "Luigi Vanvitelli", Napoli

REFERENCES:
- [Derived] Marseglia G, Licari A, Leonardi S, Papale M, Zicari AM, Schiavi L, Ciprandi G; Italian Study Group on Pediatric Allergic Rhinoconjunctivitis. A polycentric, randomized, parallel-group, study on Lertal(R), a multicomponent nutraceutical, as preventive treatment in children with allergic rhinoconjunctivitis: phase II. Ital J Pediatr. 2019 Jul 18;45(1):84. doi: 10.1186/s13052-019-0678-y. PMID 31319883

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-19): https://cdn.clinicaltrials.gov/large-docs/48/NCT03365648/Prot_SAP_000.pdf